CLINICAL TRIAL: NCT07270289
Title: Total Intravenous Anesthesia (TIVA) Versus Inhalational Anesthesia at The End of Laparoscopic Obstetric Surgery Regarding Postoperative Nausea and Vomiting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ashraf kamel, Resident doctor at Anesthesia, Intensive Care and Pain Management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tiva vs inhala anesth in ponv
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Obstetric Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients will be offed from inhalational anesthesia and Switched to propofol TIVA for the final 10 minutes of surgery
  Interventions: Procedure: inhalational anaesthesia; Procedure: total intravenous anesthesia (TIVA)
- Group B (Active Comparator): patients will be Continued on inhalational anaesthesia (sevoflurane or isoflurane per protocol)during the same final phase through extubation.
  Interventions: Procedure: inhalational anaesthesia

INTERVENTIONS:
Procedure: inhalational anaesthesia — patients will be offed from inhalational anesthesia
Procedure: total intravenous anesthesia (TIVA) — patients will be Switched Total Intravenous Anesthesia (TIVA)
  Arms: Group A

SUMMARY:
Postoperative nausea and vomiting (PONV) remain among the most common and distressing complications after general anaesthesia, with important consequences for patient comfort, satisfaction, recovery trajectories, and length of stay following surgery. The incidence of PONV is especially high after laparoscopic and gynaecological procedures due to patient- and procedure-related risk factors, making effective prevention and management a priority in perioperative care [5,8].

Anaesthetic technique is a recognized, modifiable determinant of PONV. Numerous clinical trials and randomized studies have demonstrated that the choice between propofol-based total intravenous anaesthesia (TIVA) and volatile inhalational maintenance can materially influence PONV incidence. Propofol-based TIVA has been repeatedly associated with lower rates of early and overall PONV compared with volatile agents in diverse surgical populations, supporting its role as an antiemetic strategy in addition to pharmacologic prophylaxis [1,2,4,9].

Trials specifically conducted in gynaecological and laparoscopic surgical populations report consistent reductions in nausea and vomiting with propofol maintenance compared with isoflurane or other volatile agents. These procedure-specific data are directly relevant to studies in gynecological laparoscopy, where baseline PONV risk is elevated and where anesthetic technique may yield a clinically meaningful reduction in patient morbidity [5,8,9].

Meta-analyses and systematic reviews pooling randomized controlled trials provide higher-level evidence that TIVA reduces the relative risk of PONV compared with volatile anaesthesia. Trial-sequential and pooled analyses estimate a clinically important risk reduction favoring TIVA, although effect sizes vary with study populations, prophylactic antiemetic regimens, and outcome time windows; these syntheses underpin the rationale for a targeted randomized comparison in the gynecological laparoscopic setting [2,4,10].

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-50 years.
* Elective laparoscopic procedure under general anaesthesia with endotracheal intubation.
* Expected surgical duration ≥ 30 minutes. -.Ability to consent and complete questionnaires

Exclusion Criteria:

* Pregnancy or lactation.
* BMI ≥ 40 kg/m²; severe cardiopulmonary disease; hepatic/renal failure.
* History of malignant hyperthermia or contraindication to study drugs.
* Known allergy to propofol, , , sevoflurane/desflurane.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female only
Enrollment: 98 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of post operative neasea | 24 hours
  Any episode of nausea (NRS ≥ 4/10 or requiring treatment)
incidance of postoperative vomting | 24 hours
  any episode of vomiting/retching recorded at 0-2, 2-6, and 6-24 h; need for rescue antiemetic